CLINICAL TRIAL: NCT04459000
Title: Substance Use Treatment and Access to Resources (STARS) Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STARSProj
Record Dates: First submitted 2020-06-12; First posted 2020-07-07 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Substance Use Disorders; Pregnancy Related; Child Neglect
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor/research technician will not intentionally be made aware of the participant's treatment group, although this information may not be entirely possible to prevent the tech from learning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STARs Only (Active Comparator): Consenting research participant who receive prenatal care services in the STAR clinic, but are not randomized to receive mABC home visiting services.
  Interventions: Behavioral: STARs Only
- STARS + mABC (Experimental): Consenting research participant who receive prenatal care services in the STAR clinic, and are randomized to receive mABC home visiting services.
  Interventions: Behavioral: STARS + maternal Attachment Biobehavioral Catchup home visiting model
- Control Group/CHOUM Only (No Intervention): These are research participants who were eligible to receive care in the STAR clinic, but did not opt to receive that care.

INTERVENTIONS:
Behavioral: STARS + maternal Attachment Biobehavioral Catchup home visiting model — Mothers receive up to 12 home visits from a licensed therapist focused on attachment and positive parenting in substance exposed babies. This includes 1 prenatal home visit and up to 11 postnatal visits.
  Arms: STARS + mABC
Behavioral: STARs Only — Participants receive prenatal care in the STAR clinic (a clinic specifically designed to support mothers with substance abuse who are at risk of losing their children to child welfare at birth).
  Arms: STARs Only

SUMMARY:
This study is evaluating a randomized clinical trial and a quasi-experimental observational study combined. Pregnant women with substance abuse issues are referred to the Substance Use Treatment and Recovery (STAR) prenatal clinic, and those who consent to participate in the study will be randomized to the STAR + maternal Attachment Biobehavioral Catchup (mABC) home visiting model or to the STAR only treatment group. Those who opt out of receiving prenatal care at STAR will be recruited as a control group for the QED portion. Those randomized to STAR + mABC will receive additional supports from a licensed therapist, including up to 12 home visits focused on substance exposed babies and positive parenting.

DETAILED DESCRIPTION:
This study is evaluating a randomized clinical trial and a quasi-experimental observational study combined. Pregnant women with substance abuse issues are referred to the Substance Use Treatment and Recovery (STAR) prenatal clinic, and those who consent to participate in the study will be randomized to the STAR + maternal Attachment Biobehavioral Catchup (mABC) home visiting model or to the STAR only treatment group. Those who opt out of receiving prenatal care at STAR will be recruited as a control group for the QED portion. Those randomized to STAR + mABC will receive additional supports from a licensed therapist, including up to 12 home visits focused on substance exposed babies and positive parenting. The study will focus on the following specific aims:

A. Specific Aims

The Oklahoma Department of Mental Health and Substance Abuse Services (OKDMHSAS), in partnership with two clinics at Children's Hospital at OU Medicine (CHOUM) - the Substance use Treatment And Recovery (STAR) prenatal clinic and the A Better Chance Clinic (ABCC) for infant assessment and treatment - have developed the Substance use Treatment and Access to Resources and Supports (STARS) program for pregnant women who have a substance use issue. The STARS program focuses on women residing in Oklahoma County (OK co.) who, at the time of birth, are at risk of losing their infant to state custody care (child removal). The effectiveness of combined focal services provided by the STAR (prenatal care, substance use treatment supports and postpartum care) and the ABCC (assessment, evidence-based parent training) clinics will be the target of the study described herein. The overarching goal of the study is to evaluate the impact of these services on the well-being of and permanency outcomes for children and families affected by substance abuse. The study will also evaluate the quality of service implementation and the overall project's adherence to the following objectives:

Objective 1: Develop training and cross-training to increase the knowledge base of the medical, therapy, and child welfare. The key element of this objective is to increase the state's capacity to deliver collaborative and integrated services to serve children ages 0-3 and their families. The STARS will increase the health care and child welfare workforce's capacity by disseminating emerging and evidence-based services for substance-exposed newborns and Fetal Alcohol Spectrum Disorder. The ODMHSAS and OKDHS plan to enhance cross-systems interventions that bridge agencies at policy and practice levels by pursuing procedural and policy modifications and formalize agreements to implement targeted evidence-based training that will enhance the knowledge base of statewide substance use disorder treatment providers, child welfare and health care professionals. Because of the state and local infrastructure, the ODMHSAS has developed to date, key partnerships, and access to data, the program is well-positioned to focus on substance-exposed newborns and their families as Oklahoma continues to strengthen and expand the statewide service and workforce capacity.

Objective 2: Enhance the well-being of children, parents, and families; and improve safe and permanent caregiving relationships. The key element of this objective is to improve evidence-based practices to address attachment and bonding that will serve the mother and baby. To achieve this, the STARS program will collaborate with A Better Chance Clinic (ABCC) at OUHSC to implement modified maternal Attachment Biobehavioral Catchup (mABC) adaptation for pre and postnatal babies. mABC is an intervention adapted from an evidence-based intervention for children who have experienced adversity (e.g., neglect). This adapted intervention specifically targets the challenges of infants born to opioid-dependent mothers.

Objective 3: Improve retention in substance use treatment and successful completion of treatment for parents: STARS program will utilize an array of EBPs to improve treatment retention and encourage completion of treatment services. Treatment outcomes are increased by offering services to meet the parent's needs. Motivational Interviewing (MI), Community Reinforcement Approach (CRA), and Seeking Safety (SS) and Cognitive Process Therapy for trauma (CPT) will be utilized to address the treatment needs.

Objective 4: Facilitate the implementation, delivery, and effectiveness of prevention services and programs under the Family First Prevention Services Act of 2018 for at-risk families: Under Division E, Title VII - Family First Prevention Services Act, listed under Prevention Activities under Title IV-E, it allows title IV-E dollars to fund promising, supported, and well-supported mental health and substance abuse prevention and treatment provided by a qualified clinician, and in-home parent skill-based programs, for up to 12 months for candidates for foster care and for pregnant or parenting foster youth. ODMHSAS will develop memorandums of understandings, conducting multidisciplinary teams, and providing the evidence-based services that treat families that are at risk in compliance with this services act.

Objective 5: Decrease the number of out of home placements for children by enhancing the safety of children prior to delivery: ODMHSAS with collaboration with OKDHS will develop Plans of Safe Care prior to delivery. The STARS program will implement Wraparound services to connect families to resources to support the mother and baby after delivery to ensure they have a safe environment and lifestyle.

Objective 6: Decrease the number of out of home placements for children at risk: The STARS program will provide various services and supports prior to delivery of the baby. The program will offer prenatal care; Medication-Assisted Treatment (MAT) when applicable, substance use treatment through telehealth or in-person, peer recovery, housing and employment, and aftercare supports.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman with substance abuse issue occurring during pregnancy
* Eligible for services at the STAR prenatal clinic
* Speaks/comprehends English

Exclusion Criteria:

* Unable to read English at 8th grade comprehension level
* Those outside of Oklahoma City metropolitan area.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 242 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Mother substance use | Change from baseline to 18 months post birth of child
  Are there group differences in the rate of mother's substance use? Substance use measured using Addiction Severity Index (ASI) assessment self-report. Frequencies of use of different drugs will be monitored.
Mother contraceptive use | Change from baseline to 18 months post birth of child
  Are there group differences in the rate of mother's contraceptive use? Substance use measured using risk and contraception items from Youth Risk Behavior Surveillance System survey. Frequencies will be monitored for change.
Mother depressive symptoms | Change from baseline to 18 months post birth of child
  Center for Epidemiological Studies Depression Screener score
Child development | Change from baseline to 18 months post birth of child
  Infant and Toddler Sensory Profile
Child development | Change from baseline to 18 months post birth of child
  Bayley Scales
Child welfare involvement | Change from baseline to 18 months post birth of child
  Are there group differences in the rate of child removals by protective services? Count of children removed using Child Welfare data.
Child welfare reunifications | Change from baseline to 18 months post birth of child
  Are there group differences in the rate of child reunifications among participants who lose temporary custody at birth? Count of reunifications for those who lost custody at birth based on child welfare data.

CONTACTS AND LOCATIONS:
Overall Officials: David Bard, PhD, Principal Investigator — OUHSC
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No